CLINICAL TRIAL: NCT05658159
Title: Physiological and Dietary Characteristics of Boys and Girls High School Basketball Players
Status: Completed | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2202
Record Dates: First submitted 2022-12-09; First posted 2022-12-20 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Bone Health
Keywords: bone health; high school; diet; basketball; vitamin D; DXA; DEXA; nutrition; diet quality; energy intake
MeSH Terms: interventions — Vitamin D Response Element; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vitamin D Assessment: ZRT Laboratories, Beaverton, OR. A finger stick will be used to obtain a capillary blood sample for assessment of Vitamin D (25(OH)D)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vitamin D — Finger stick capillary blood sampling using test from ZRT Laboratories, Beaverton, OR
  Other Names: Vitamin D (25(OH)D)
Diagnostic Test: DXA scan — 10 minute scan using scanner by GE Lunar, Madison, WI
  Other Names: Dual Xray Absorptiometry
Other: Nutrition analysis — Analysis of 24-h recalls will be conducted by a registered dietician using Nutritionist Pro software by Axxya Systems, Redmond, WA

SUMMARY:
In a population of boys and girls high school basketball players, the primary objectives are to assess 1) bone mineral density and vitamin D status, and 2) energy intake and dietary quality.

The secondary objectives are to assess 1) nutrients related to bone health (calcium, magnesium, vitamin K, protein) and 2) protein intake over the day.

Data collection takes place pre-, mid-, and post-season.

DETAILED DESCRIPTION:
This study will assess the dietary intake male and female 14-19 year old student athletes, specifically energy intake and dietary quality (i.e. how closely do their diets meet recommendations).

Investigators hypothesize that vitamin D status will be suboptimal in most participants though bone density will be normal.

Investigators hypothesize that participants will maintain energy balance over the course of the season (no significant changes to body mass or body composition) but dietary quality will not meet recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males between the ages of 14-19 years old.
2. Non-smoker
3. Currently enrolled in the IMG basketball program.
4. Willing to fast overnight prior to testing.
5. Willing to do a finger stick for the Vitamin D assessment.
6. Able to give verbal and written informed consent for participation as well as obtain parental consent if <18 years of age.
7. If an athlete would like to participate but English is not their first language, we will liaise with an interpreter on the IMG campus to inform him / her of the study protocol and procedures.

Exclusion Criteria:

1. Expulsion from school for any reason.
2. Leaving the IMG basketball program.
3. Pregnant or planning to become pregnant

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Male and female high school basketball players
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Normal whole body bone density would be better.
  whole body
Bone mineral density | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Normal spine bone density would be better.
  spine
Bone mineral density | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Normal total hip bone density would be better.
  total hip
Bone mineral density | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Normal femoral neck bone density would be better.
  femoral neck
Bone mineral density | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Adequacy will be defined as a value > 32 ng/mL. Higher Vitamin D values would be better.
  vitamin D status
Energy intake | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Energy intake that meets recommendations would be better.
  24 hour recall
Dietary quality | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Diet quality that meets recommendations would be better.
  24 hour recall

SECONDARY OUTCOMES:
Assess nutrients related to bone health (calcium) | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Calcium intake that meets recommendations would be better.
  Calcium intake via 24 hour recall and calcium supplement, if any
Assess nutrients related to bone health (magnesium) | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Magnesium intake that meets recommendations would be better.
  Magnesium intake via 24 hour recall and magnesium supplement, if any
Assess nutrients related to bone health (vitamin K) | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Vitamin K intake that meets recommendations would be better.
  Vitamin K intake via 24 hour recall and vitamin K supplement, if any
Assess nutrients related to bone health (protein) | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Protein intake that meets recommendations would be better.
  Protein intake via 24 hour recall
Protein intake over the day | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Looking at pattern of protein intake.
  Times of day protein is consumed

OTHER OUTCOMES:
Assess frequency of consuming carbohydrate during training | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Looking at pattern of carbohydrate intake.
  Carbohydrate intake via 24 hour recall
Assess current intake of supplements | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023) in consumption of supplements. Better or worse outcome not applicable.
  Measure intake of supplements (pills, powders, gummies, etc.) via 24 hour recall and reported concomitant meds/supplements
Weight | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). No desired direction of change, expecting it to remain contstant.
  Body weight scale accuracy to one tenth of a kilogram using a scale from data Weighing Systems, Wood Dale, IL
Height | Changes from basketball pre-season (October 2022) to mid-season (January 2023) to post-season (April 2023). Better or worse direction not applicable.
  Participants standing and seated height will be measured by electronic stadiometry to the nearest cm using QuickMedical stadiometer, Warwick, RI

CONTACTS AND LOCATIONS:
Overall Officials: Kris Osterberg, PhD,RD,CSSD, Principal Investigator — PepsiCo, Inc. Sports Science
Locations (1):
- IMG Academy, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No